CLINICAL TRIAL: NCT07255781
Title: Shared Mechanisms Contributing to Non-Alcoholic Fatty Liver Disease (NAFLD) and Psoriatic Disease (PD) Severity With Guselkumab Therapy [EMERGE]
Brief Title: Shared Pathways Between Non-Alcoholic Fatty Liver Disease and Psoriatic Disease With Guselekumab Therapy
Acronym: EMERGE
Status: Not yet recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Monica Guma, Associate Professor, University of California, San Diego
Other Study IDs: CNTO1959PSA4014
Record Dates: First submitted 2025-09-24; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Psoriasis (PsO); PsA (Psoriatic Arthritis); NAFLD (Nonalcoholic Fatty Liver Disease)
Keywords: psoriasis; psoriatic arthritis; guselkumab; NAFLD; non-alcoholic fatty liver disease
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic; Non-alcoholic Fatty Liver Disease | interventions — guselkumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Active Psoriatic Disease: Patients with active psoriatic disease (diagnosed with psoriasis and/or psoriatic arthritis) who are planning to start Guselkumab as part of their standard of care.
  Interventions: Drug: Guselkumab Prefilled Syringe [Tremfya]

INTERVENTIONS:
Drug: Guselkumab Prefilled Syringe [Tremfya] — This trial aims to recruit patients who have psoriatic disease, have evidence of fatty liver disease, and have a BMI over 25, who are planning to start Guselkumab(Tremfya) as recommended by their primary rheumatologist or dermatologist

SUMMARY:
The goal of this research study is to better understand if there is an association between non-alcoholic fatty liver disease (NAFLD) and active psoriatic disease (PD), and to assess the effect of Guselkumab (a medication approved by the FDA instead of the standard of care to treat PD), for NAFLD patients who receive Guselkumab for their PD.

DETAILED DESCRIPTION:
This observational research study aims to provide information on the mechanisms behind the transition from NAFLD to high-risk NASH in the PD population. Overlapping mechanisms of disease in NAFLD and PD may account for increased disease prevalence and severity, and shared drivers of disease progression offer the opportunity to ameliorate both disease entities by targeting a single pathway. This is a longitudinal study that requires two visits from individuals with psoriatic disease. Subjects must have NAFLD and at least one criterion for active psoriatic disease: i) at least 1 swollen joint or 1 site of active enthesitis; and/or (ii at least 1 psoriatic plaque to qualify for the study. The aim of the study is to determine the effect of biological therapies in liver disorders in patients with PD, in addition to the effect on joint and skin manifestations.

ELIGIBILITY:
Inclusion criteria:

* Adults with a diagnosis of PsA fulfilling the classification for PsA (CASPAR) criteria.
* Overweight or obese by BMI ≥ 25.0 kg/m2 or ≥ 23.0 for Asian participants
* Patients are starting Guselkumab therapy as indicated by primary rheumatologist
* Elevated liver fat on controlled attenuation parameter (CAP) ≥ 288 dB/m, which is consistent with NAFLD after exclusion of secondary causes of liver disease8.

Exclusion Criteria:

* Evidence of other causes of chronic liver disease
* Hepatitis B as defined as presence of hepatitis B surface antigen (HBsAg).
* Previous or current infection with Hepatitis C as defined by presence of hepatitis C virus Ab in serum (anti-HCV Ab).
* Autoimmune hepatitis as defined by anti-nuclear antibody (ANA) of 1:160 or greater and liver histology consistent with autoimmune hepatitis or previous response to immunosuppressive therapy.
* Autoimmune cholestatic liver disorders as defined by elevation of alkaline phosphatase and anti-mitochondrial antibody of greater than 1:80 or liver histology consistent with primary biliary cirrhosis or elevation of alkaline phosphatase and liver histology consistent with sclerosing cholangitis.
* Wilson disease as defined by ceruloplasmin below the limits of normal and liver histology consistent with Wilson disease.
* Alpha-1-antitrypsin deficiency as defined by alpha-1-antitrypsin level less than normal and liver histology consistent with alpha-1-antitrypsin deficiency.
* Hemochromatosis as defined by presence of 3+ or 4+ stainable iron on liver biopsy and homozygosity for C282Y or compound heterozygosity for C282Y/H63D.
* Drug-induced liver disease as defined on the basis of typical exposure and history.
* Bile duct obstruction as shown by imaging studies.
* History of gastrointestinal bypass surgery or ingestion of medications known to produce steatosis, such as corticosteroids, high-dose estrogen, tamoxifen, amiodarone, or tetracycline in the previous 6 months.
* Evidence of cirrhosis or previously known cirrhosis based on the results from a previous liver biopsy or history of portal hypertension presented by ascites, hepatic encephalopathy, or varices
* Presence of regular and/or excessive use of alcohol (defined as >30g/day for males and >15g/day for females) for a period longer than 2 years at any time in the last 10 years
* The subject is a pregnant or nursing female
* History of known HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total sample of approximately 20 PD patients from UCSD rheumatology clinics. 50% of patients screened will meet the inclusion criteria for NAFLD. To provide equal representation of the Psoriatic Disease population, 10 patients who meet the inclusion criteria for moderate to severe plaque psoriasis, and approximately 10 patients who meet the inclusion criteria for active psoriatic arthritis, will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in NAFLD severity | 6 months
  Improvement of NAFLD severity is defined by MRI-PDFF responders (relative decline in liver fat ≥30%) vs non-responders (relative decline in liver fat <30%) at Week 24

SECONDARY OUTCOMES:
Improvement in skin psoriasis severity as defined by PASI90 (Psoriasis Area and Severity Index) response | 6 months
Improvement in joint arthritis as defined by an improvement of ≥ 5 of DAPSA (Disease Activity in Psoriatic Arthritis) | 6 months
17 units per liter improvement in alanine aminotransferase(ALT) in those patients with elevated ALT at baseline. | 6 months
  Elevated ALT is defined as ≥ 30 U/L.